CLINICAL TRIAL: NCT06077175
Title: EFFECT of HAND MASSAGE on PATIENTS AFTER ACUTE CORONARY SYNDROME on the COMFORT and ANXIETY LEVEL
Brief Title: HAND MASSAGE AFTER ACUTE CORONARY SYNDROME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem Ceyhan, Teaching staff, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AKSHAND
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2023-10

CONDITIONS: Acute Coronary Syndrome; Anxiety
Keywords: acute coronary syndrome; anxiety; comfort; han massage
MeSH Terms: conditions — Acute Coronary Syndrome; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: hand massage group
- Control group (No Intervention)

INTERVENTIONS:
Other: hand massage group — Each individual will receive a 10-minute hand massage, 5 minutes for each hand. Since the speed and number of repetitions of the massage movements should be at normal frequency, the massage will be performed at a speed that does not disturb the individual, is not stimulating and has a calming effect, and will not tire the practitioner. In the massage, effleurage (stroking) and friction (circular rubbing) movements will be used, which have a circulation-supporting and tissue-relaxing effect. Evaluations will be made within 30 minutes after the hand massage.
  Arms: intervention group

SUMMARY:
Patients suffering from Acute coronary syndrome may be hospitalized again in a shorter time than expected, and after being discharged, they may live within the limitations imposed by the disease until the end of their lives. This situation causes anxiety in individuals. Today, various methods are used to reduce high levels of anxiety. Massage is the planned and purposeful application of touch and is the most common, most important and oldest complementary treatment used in traditional practices. It is also thought that the comfort levels of individuals experiencing ACS will increase by reducing their anxiety. This study was planned to determine the effect of hand massage applied to patients with ACS on comfort, anxiety level and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing Acute Coronary Syndrome for the first time,
* Anxiety score of 16 and above (moderate and severe anxiety)
* 18 years and above,
* No psychiatric disease,
* Patients who do not have communication problems and are competent to answer all questions,

Exclusion Criteria:

* Patients with uncontrolled Diabetes mellitus
* Patients who cannot communicate and have confusion,
* Those who have any limb, vascular problem or wound that prevents hand massage,
* Thrombophlebitis, occlusive arterial disease, fever etc. Those for whom massage therapy is inconvenient due to illness,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Scale | It will be done before the massage application, 24 hours after arrival in the intensive care unit.
  It is a self-rating scale used to determine the frequency of anxiety symptoms experienced by individuals.
Beck Anxiety Scale | It will be applied on the 4th day at the end of the application.
  It is a self-rating scale used to determine the frequency of anxiety symptoms experienced by individuals.

SECONDARY OUTCOMES:
General Comfort Scale | It will be done before the massage application, 24 hours after arrival in the intensive care unit.
  It is used to determine the comfort level of patients.
General Comfort Scale | It will be applied on the 4th day at the end of the application.
  It is used to determine the comfort level of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mei L, Miao X, Chen H, Huang X, Zheng G. Effectiveness of Chinese Hand Massage on Anxiety Among Patients Awaiting Coronary Angiography: A Randomized Controlled Trial. J Cardiovasc Nurs. 2017 Mar/Apr;32(2):196-203. doi: 10.1097/JCN.0000000000000309. PMID 26646596
- [Background] Alimohammad HS, Ghasemi Z, Shahriar S, Morteza S, Arsalan K. Effect of hand and foot surface stroke massage on anxiety and vital signs in patients with acute coronary syndrome: A randomized clinical trial. Complement Ther Clin Pract. 2018 May;31:126-131. doi: 10.1016/j.ctcp.2018.01.012. Epub 2018 Feb 13. PMID 29705444
- [Background] Cavdar AU, Yilmaz E, Baydur H. The Effect of Hand Massage Before Cataract Surgery on Patient Anxiety and Comfort: A Randomized Controlled Study. J Perianesth Nurs. 2020 Feb;35(1):54-59. doi: 10.1016/j.jopan.2019.06.012. Epub 2019 Sep 21. PMID 31551136
- [Background] Kunikata H, Watanabe K, Miyoshi M, Tanioka T. The effects measurement of hand massage by the autonomic activity and psychological indicators. J Med Invest. 2012;59(1-2):206-12. doi: 10.2152/jmi.59.206. PMID 22450009